CLINICAL TRIAL: NCT04772703
Title: DNA Damage in Critically Ill Patients With SARS-CoV-2 Infection With Organ Failure
Brief Title: DNA Damage in Critically Ill COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Sponsor
Other Study IDs: CVV_COVID-19_DNA
Record Dates: First submitted 2021-02-25; First posted 2021-02-26 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Covid19; Organ Failure, Multiple; DNA Damage
MeSH Terms: conditions — COVID-19; Multiple Organ Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: COMET ASSAY — The description in the detailed description of the study

SUMMARY:
Critically ill patients with COVID-19 are exposed to high oxidative stress which is potential harm to the DNA. Peripheral lymphocytes' DNA will be investigated using the comet assay on changes in oxidative damage to the purine and pyrimidine bases and single-stranded DNA breaks.

DETAILED DESCRIPTION:
Data from hospital documentation will be recorded for all patients: demographic data, clinical data (Horowitz index, the necessity of pronation position, opening maneuvers, connection to ECMO, state of the circulation and other organ functions), laboratory data: parameters of inflammatory activity and COVID-19 specific markers (blood count with differential leukocyte count, CRP, IL-6, ferritin, procalcitonin, D-dimers).

In the study, 4 ml of heparinized peripheral blood will be collected for analytical purposes beyond standard practice for lymphocyte isolation and monitoring of oxidative DNA damage upon admission to the ICU (D1), after 2 days (D3) and on day 7 (D7) of the hospitalization. The same blood sample will be used to determine EPA and DHA omega-3 in erythrocyte membranes. At the same intervals and frequency, 10 ml of urine will be collected for the determination of 8-hydroxy-2-deoxyquanosine (8-OHdG), so a total of 30 ml of urine will be collected for analytical purposes.

Details for analytical processing: peripheral blood lymphocyte damage will be assessed using the alkaline COMET ASSAY method for DNA breakage and modified COMET ASSAY using specific enzymes for the detection of oxidized bases, endonuclease III (ENDO III) for the detection of oxidized pyrimidines and formamidopyrimidine DNA glycosylase (FPG) for the detection of oxidized purines. Leukocyte repair capacity will be determined using a modified COMET ASSAY, which uses extracts of patient lymphocytes and HeLa cells with defined DNA damage. The extent of 8-hydroxy-2-deoxyquanosine (8-OHdG) DNA damage in patients' urine will be determined by determining the concentration of 8-OHdG by ELISA.

ELIGIBILITY:
Inclusion Criteria:

* critically ill adult patient admitted to ICU with positive RT-PCR test or bed-side antigen test on COVID-19 with signs and symptoms of organ failure
* informed consent

Exclusion Criteria:

* rejection by the patient to sign an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients admitted to ICU with signs and symptoms of organ failure, mainly respiratory failure. Need for means of respiratory and/or circulatory support. A positive test of COVID-19: RT-PCR test or bed-side antigen test.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
single-stranded DNA breaks | One week
  Changes in the single-stranded DNA breaks in peripheral lymphocytes
oxidation of DNA bases | One week
  Changes in oxidised purine and pyrimidine bases of peripheral lymphocytes DNA

SECONDARY OUTCOMES:
Mortality | One month
  All cause 30-day mortality

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Hradec Kralove, Hradec Králové, Třebeš, Czechia

IPD SHARING:
Plan to Share IPD: No